CLINICAL TRIAL: NCT04013698
Title: Effects of Chest Wall and Lung Elastances on Intracranial Pressure and Brain-specific Multimodal Monitoring in Ventilated Brain Injured Patients
Brief Title: Influence of Respiratory Mechanics on Brain-specific Monitoring in Brain-injured Patients
Acronym: ABIVENT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the COVID epidemics, starting with patient recruitement was not possible.
Sponsor: Piquilloud Imboden Lise (Other)
Responsible Party: Sponsor-Investigator, Piquilloud Imboden Lise, Sponsor-Investigator, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ABIVENT
Record Dates: First submitted 2019-07-01; First posted 2019-07-10 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2020-11

CONDITIONS: Brain Injuries
Keywords: ventilation; brain injuries; PEEP; esophageal pressure
MeSH Terms: conditions — Brain Injuries; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Patients included will receive volume assist-control ventilation with PEEP set at 5 cmH2O and 15 cmH2O in a randomized order (crossover design). Each setting will be applied during 45 minutes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEP level 5 cmH2O to 15 cmH2O (Experimental)
  Interventions: Other: PEEP level 5 cmH2O; Other: PEEP level 15 cmH2O
- PEEP level 15 cmH2O to 5 cmH2O (Experimental)
  Interventions: Other: PEEP level 5 cmH2O; Other: PEEP level 15 cmH2O

INTERVENTIONS:
Other: PEEP level 5 cmH2O — PEEP level set for 45 minutes
Other: PEEP level 15 cmH2O — PEEP level set for 45 minutes

SUMMARY:
Increase in intracranial pressure (ICP) could be associated with increase in positive end-expiratory pressure (PEEP) level. Data are however disparate and interactions between ventilation with high PEEP and intracranial circulation are still debated. Individual patient's chest wall elastance could have a key role in determining the effects of PEEP on ICP, since it dictates which proportion of the applied PEEP is transmitted to the pleural space, thus increasing central venous pressure (CVP) and reducing cerebral venous return. Measurement of esophageal pressure with a dedicated probe allows partitioning of respiratory system elastance into its lung and chest wall components, thus permitting to study this phenomenon. Multimodal intracranial monitoring permits to study the effects of PEEP on more advanced brain-specific indices such as brain tissue oxygen (PtiO2), cerebral microdialysis data, transcranial doppler ultrasound-derived flow measurements and automated pupillometry, besides ICP.

This study aims to test the association between the ratio of chest wall to respiratory system elastance and PEEP-induced variations in ICP and brain-specific multimodal monitoring indices. This study will evaluate the relative role of other selected measures of respiratory mechanics, hemodynamic variables and intracranial compliance, in order to establish the role of individual respiratory mechanics in the interplay of physiological factors affecting the effects of positive pressure ventilation on the brain.

Patients will undergo two periods of ventilation at two different levels of PEEP (5 and 15 cmH2O) in a randomized cross-over order. At the end of each period, cardiorespiratory clinical data, ICP and other advanced multimodal neuromonitoring data (brain tissue oxygen tension, cerebral microdyalisis analytes, transcranial doppler ultrasound and automated infrared pupillometry data) will be collected. Systematic respiratory mechanics assessment (including calculation of chest wall and lung elastances and estimation of the amount of recruitment versus overdistension due to PEEP by means of a single-breath derecruitment trial), echocardiography and arterial blood gas analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Acute brain injury of any etiology requiring multimodal brain monitoring (intraparenchymal intracranial pressure, brain-tissue oxygen tension and cerebral microdialysis)
* Controlled mechanical ventilation via endotracheal tube
* Patient needing deep sedation

Exclusion Criteria:

* pregnancy
* contraindications to nasogastric probe placement: basilar skull or significant naso-facial fractures, significant esophageal or gastric trauma or bleeding, previous esophageal surgery, significant bleeding diathesis (spontaneous aPTT > 60 sec, PT < 40%, INR > 1.8, platelets < 50000/mm3), known esophageal or gastric varices
* decompressive craniectomy
* intracranial pressure monitoring method other than intraparenchymal (e.g. connected to external ventricular drain)
* severe relevant physiological instability contraindicating an increase in PEEP: severe baseline intracranial pressure elevation (> 20 mmHg), severe hemodynamic instability (defined as norepinephrine requirements > 0.5 μg/kg/min or cardiogenic shock, defined as any use of dobutamine)
* conditions that interfere with accurate measurements of respiratory mechanics: bronchopleural fistula, pneumothorax.
* Withhold of life-sustaining therapy for medical reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Correlation between Ers/Ecw and change in ICP between the two PEEP levels | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Respiratory mechanics; intracranial pressure monitoring
  Ers/Ecw = chest wall to respiratory system elastances ratio; ICP = intracranial pressure

SECONDARY OUTCOMES:
Correlation between Ecw/Ers and the following neuromonitoring indices at the two PEEP levels: PtiO2, LPR, NPI; MFV, DFV and PI. | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Respiratory mechanics; brain tissue oxygen tension; cerebral microdyalisis analytes; automated infrared pupillometry; transcranial doppler ultrasound
  Ers/Ecw = chest wall to respiratory system elastances ratio; PtiO2 = brain tissue oxygen tension; LPR = lactate/pyruvate ratio; NPI = neurological pupil index; MFV = mean flow velocity; DFV = diastolic flow velocity; PI = pulsatility index
Effect of the two different levels of PEEP on NPI. | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Automated infrared pupillometry
  NPI = neurological pupil index
  PtiO2 = brain tissue oxygen tension; LPR = lactate/pyruvate ratio; NPI = neurological pupil index
Effect of the two different levels of PEEP on the following transcranial doppler ultrasound variables: MFV, DFV and PI. | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Transcranial doppler ultrasound
  MFV = mean flow velocity; DFV = diastolic flow velocity; PI = pulsatility index
Effect of the two different levels of PEEP on LPR. | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Cerebral microdyalisis analytes
  LPR = lactate/pyruvate ratio
Effect of the two different levels of PEEP on PtiO2. | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Brain tissue oxygen tension.
  PtiO2 = brain tissue oxygen tension
Effect of the two different levels of PEEP on the following intravascular pressures: CVP, MAP, CPP. | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Invasive intravascular pressures.
  CVP = central venous pressure; MAP = mean arterial pressure; CPP = cerebral perfusion pressure
Effect of the two different levels of PEEP on the following echocardiographic measurements: LVOT VTI, CO. | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Echocardiography.
  LVOT VTI = left ventricle outflow tract velocity-time integral; CO = cardiac output (echocardiographically estimated).
Effect of the two different levels of PEEP on the dose of vasopressors/inotropes and volume of fluid boluses administered. | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Administered drugs and fluids.
Correlation between Ers/Ecw and the following parameters at the two PEEP levels: LVOT VTI, CO; CVP, MAP, CPP; dose of vasopressors/inotropes and volume of fluid boluses administered. | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Respiratory mechanics; echocardiography; invasive intravascular pressures; administered drugs and fluids
  LVOT VTI = left ventricle outflow tract velocity-time integral; CO = cardiac output (echocardiographically estimated); CVP = central venous pressure; MAP = mean arterial pressure; CPP = cerebral perfusion pressure
Correlation between Pes_end-exp and the following parameters at the two PEEP levels: ICP, PtiO2, LPR, NPI, MFV, DFV, PI; CVP, MAP, CPP, LVOT VTI, CO, dose of vasopressors/inotropes and volume of fluid boluses administered. | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Respiratory mechanics; intracranial pressure monitoring, Brain tissue oxygen tension; cerebral microdyalisis analytes; automated infrared pupillometry; transcranial doppler ultrasound; Echocardiography; invasive intravascular pressures; administered drugs and fluids.
  ICP = intracranial pressure; PtiO2 = brain tissue oxygen tension; LPR = lactate/pyruvate ratio; NPI = neurological pupil index; MFV = mean flow velocity; DFV = diastolic flow velocity; PI = pulsatility index; CVP = central venous pressure; MAP = mean arterial pressure; CPP = cerebral perfusion pressure; LVOT VTI = left ventricle outflow tract velocity-time integral; CO = cardiac output (echocardiographically estimated)
Correlation between Rec/PEEPvol and the following parameters at the two PEEP levels: ICP, PtiO2, LPR, NPI, MFV, DFV, PI; CVP, MAP, CPP, LVOT VTI, CO, dose of vasopressors/inotropes and volume of fluid boluses administered. | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Respiratory mechanics; intracranial pressure monitoring, Brain tissue oxygen tension; cerebral microdyalisis analytes; automated infrared pupillometry; transcranial doppler ultrasound; Echocardiography; invasive intravascular pressures; administered drugs and fluids.
  Rec/PEEPvol = recruited volume to PEEP-related volume ratio; ICP = intracranial pressure; PtiO2 = brain tissue oxygen tension; LPR = lactate/pyruvate ratio; NPI = neurological pupil index; MFV = mean flow velocity; DFV = diastolic flow velocity; PI = pulsatility index; CVP = central venous pressure; MAP = mean arterial pressure; CPP = cerebral perfusion pressure; LVOT VTI = left ventricle outflow tract velocity-time integral; CO = cardiac output (echocardiographically estimated)
Correlation between Vd/Vt and the following parameters at the two PEEP levels: ICP, PtiO2, LPR, NPI, MFV, DFV, PI; CPP | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Respiratory mechanics; intracranial pressure monitoring, brain tissue oxygen tension; cerebral microdyalisis analytes; automated infrared pupillometry; transcranial doppler ultrasound; invasive intravascular pressures.
  Vd/Vt = dead space to tidal volume ratio; ICP = intracranial pressure; PtiO2 = brain tissue oxygen tension; LPR = lactate/pyruvate ratio; NPI = neurological pupil index; MFV = mean flow velocity; DFV = diastolic flow velocity; PI = pulsatility index; CVP = central venous pressure; CPP = cerebral perfusion pressure
Correlation between baseline PI at transcranial doppler ultrasound and the following parameters at the two PEEP levels: ICP, PtiO2, LPR, NPI, MFV, DFV, PI; LVOT VTI, CO, MAP, CPP. | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Intracranial pressure monitoring, Brain tissue oxygen tension; cerebral microdyalisis analytes; automated infrared pupillometry; transcranial doppler ultrasound; Echocardiography; invasive intravascular pressures.
  PI = pulsatility index; ICP = intracranial pressure; PtiO2 = brain tissue oxygen tension; LPR = lactate/pyruvate ratio; NPI = neurological pupil index; MFV = mean flow velocity; DFV = diastolic flow velocity; PI = pulsatility index; LVOT VTI = left ventricle outflow tract velocity-time integral; CO = cardiac output (echocardiographically estimated); MAP = mean arterial pressure; CPP = cerebral perfusion pressure
Correlation between CVP and the following parameters at the two PEEP levels : ICP, PtiO2, LPR, NPI, MFV, DFV, PI; LVOT VTI, CO, MAP, CPP, dose of vasopressors/inotropes and volume of fluid boluses administered. | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Intracranial pressure monitoring, Brain tissue oxygen tension; cerebral microdyalisis analytes; automated infrared pupillometry; transcranial doppler ultrasound; Echocardiography; invasive intravascular pressures; administered drugs and fluids.
  CVP = central venous pressure; ICP = intracranial pressure; PtiO2 = brain tissue oxygen tension; LPR = lactate/pyruvate ratio; NPI = neurological pupil index; MFV = mean flow velocity; DFV = diastolic flow velocity; PI = pulsatility index; LVOT VTI = left ventricle outflow tract velocity-time integral; CO = cardiac output (echocardiographically estimated); MAP = mean arterial pressure; CPP = cerebral perfusion pressure
Correlation between LVOT VTI and the following parameters at the two PEEP levels: PtiO2, LPR, NPI, MFV, DFV, PI; MAP, CPP, dose of vasopressors/inotropes and volume of fluid boluses administered. | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Brain tissue oxygen tension; cerebral microdyalisis analytes; automated infrared pupillometry; transcranial doppler ultrasound; echocardiography, invasive intravascular pressures; administered drugs and fluids.
  LVOT VTI = left ventricle outflow tract velocity-time integral; PtiO2 = brain tissue oxygen tension; LPR = lactate/pyruvate ratio; NPI = neurological pupil index; MFV = mean flow velocity; DFV = diastolic flow velocity; PI = pulsatility index; MAP = mean arterial pressure; CPP = cerebral perfusion pressure
Correlation between PtiO2 and the following parameters at the two PEEP levels: ICP, MAP, dose of vasopressors/inotropes and volume of fluid boluses administered. | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Intracranial pressure monitoring, brain tissue oxygen tension; invasive intravascular pressures; administered drugs and fluids.
  PtiO2 = brain tissue oxygen tension; ICP = intracranial pressure; MAP = mean arterial pressure
Correlation between LPR and the following parameters at the two PEEP levels: ICP, MAP, dose of vasopressors/inotropes and volume of fluid boluses administered. | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Intracranial pressure monitoring, cerebral microdyalisis analytes; invasive intravascular pressures; administered drugs and fluids.
  LPR = lactate/pyruvate ratio; ICP = intracranial pressure; MAP = mean arterial pressure
Correlation between NPI and the following parameters at the two PEEP levels: ICP, MAP, dose of vasopressors/inotropes and volume of fluid boluses administered. | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Intracranial pressure monitoring, automated infrared pupillometry; invasive intravascular pressures; administered drugs and fluids.
  NPI = neurological pupil index; ICP = intracranial pressure; MAP = mean arterial pressure
Correlation between doppler indices (MFV, DFV and PI) and the following parameters at the two PEEP levels: ICP, MAP, dose of vasopressors/inotropes and volume of fluid boluses administered. | Recorded every minute during 10 minutes at the end of each 45-minute period (PEEP 5 and 15 cmH2O), 90 minutes
  Intracranial pressure monitoring, transcranial doppler ultrasound; invasive intravascular pressures; administered drugs and fluids.
  MFV = mean flow velocity; DFV = diastolic flow velocity; PI = pulsatility index; ICP = intracranial pressure; MAP = mean arterial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Lise Piquilloud, MER&PD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Lausanne University Hospitals, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided